CLINICAL TRIAL: NCT04347759
Title: Symptom Care at Home-Heart Failure: Developing and Piloting a Symptom Monitoring and Self-Management Coaching System for Patients With Heart Failure
Brief Title: Symptom Care at Home-Heart Failure
Acronym: SCH-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Utah (Other)
Responsible Party: Principal Investigator, Youjeong Kang, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00007523; K23HL148545 (NIH)
Record Dates: First submitted 2020-04-01; First posted 2020-04-15 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure; Symptoms and Signs
Keywords: Symptom Management; Technology
MeSH Terms: conditions — Heart Failure; Signs and Symptoms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symptom Care at Home with Coaching Messages (Experimental): Participants randomized to automated daily monitoring and real-time self-management coaching.
  Interventions: Behavioral: Coaching Messages; Behavioral: Automated Daily Monitoring
- Usual Care (Active Comparator): Participants randomized to automated daily monitoring only.
  Interventions: Behavioral: Automated Daily Monitoring

INTERVENTIONS:
Behavioral: Coaching Messages — Participants receive real-time self-management coaching messages based on the severity of their symptoms. When participants call, the IVR system will ask them about each of the selected symptoms, and the patient will report symptom presence and severity numerically with the touchtone keypad.
  Arms: Symptom Care at Home with Coaching Messages
Behavioral: Automated Daily Monitoring — Participants report daily symptoms and symptom severity. There are three categories of severity based on a numeric scale of 1 to 3 for mild symptoms, 4 to 7 for moderate symptoms, and 8 to 10 for severe symptoms.

SUMMARY:
This project aims to adapt a computer-interface telephonic interactive voice response system that monitors symptoms and provides real-time, self-management coaching messages based on heart failure patient-reported outcomes.

DETAILED DESCRIPTION:
Keeping heart failure (HF) patients at home with a low symptom burden after hospital discharge is challenging. HF patients may suffer worsening symptoms over time without seeking medical advice leading to poor quality of life and readmission to the hospital. Evidence shows that delay in HF symptom recognition and poor self-management are associated with unplanned HF-related emergency department (ED) visits and rehospitalizations. Clinical trials aimed at preventing rehospitalization using telemonitoring of physical changes, such as daily weights, have shown limited utility.

Understanding patients' experiences of HF symptoms and engagement in appropriate self-management are key to maintaining disease stability. Cancer studies have shown that symptom burden can be effectively decreased using automated home monitoring and self-management coaching. A recent cancer study has demonstrated that patients receiving cancer chemotherapy achieved a 40% reduction in symptoms using Symptom Care at Home (SCH), a telephone-computer interface interactive voice response (IVR) system pairing patient-reported symptoms with automated real-time self-management coaching. While a few HF studies have used interventions that monitored symptoms, no studies have tested a system that monitors and provides real-time self-management coaching tailored to specific patient-reported outcomes (PRO). The objective of this study is to adapt the SCH system to HF and conduct a pilot randomized controlled trial (RCT) to assess the feasibility, acceptability, and preliminary efficacy of the Symptom Care at Home - Heart Failure (SCH-HF) system.

Participants are randomized to receive usual care consisting of automated daily monitoring, or to receive the intervention, which includes automated daily monitoring and real-time self-management coaching.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of heart failure
* New York Heart Association (NYHA) Classification of the Stages of Heart Failure Class I - IV
* Ability to read, understand, and speak in English
* Will be discharged home
* Has daily access to any type of telephone

Exclusion Criteria:

* A score of 0 or 1-2 with an abnormally drawn clock on the Mini-Cog
* Discharged home on hospice care
* End-stage renal failure
* Wait list for heart transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Self-Care of Heart Failure Index (SCHFI) Score | Baseline (at the time of hospital discharge, pre-intervention), Day 30 (post-intervention)
  The Self-Care of Heart Failure Index, version 7.2, is a 29-item instrument with separate scales assessing self-care maintenance, symptom perception, and self-care management. Responses to items are given on a 5-point scale. Scores for each of the three scales are summed and standardized with scores ranging from 0 to 100. Higher scores indicate better self-care, with scores of 70 or higher indicating adequate levels of heart failure self-care.

SECONDARY OUTCOMES:
Number of Participants Re-hospitalized | Up to 30 days after hospital discharge
  The re-hospitalization rate will be examined between study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Youjeong Kang, PhD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - University of Utah Health, Salt Lake City, Utah